CLINICAL TRIAL: NCT07104916
Title: A Pilot Mechanistic RCT of Psilocybin With Mindfulness-based Therapy vs Support for Posttraumatic Stress Disorder (PTSD)
Brief Title: Mindfulness-based Psilocybin Therapy for PTSD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anthony P King (Other)
Responsible Party: Sponsor-Investigator, Anthony P King, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20250273
Record Dates: First submitted 2025-07-28; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder; Depression - Major Depressive Disorder
Keywords: Psychedelic; functional MRI; Mindfulness-based Cognitive Therapy; Psilocybin; microstructural neuroplasticity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This is a Phase II, randomized, assessor-blind study in participants with PTSD. The study will investigate the changes in brain activity, connectivity, and microstructural neuroplasticity assessed using EEG/EMG and fMRI / DWI measures after administration of one oral dose of psilocybin, accompanied either with standard "psychological support" or with active therapy called MBCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin with support + MBCT (Experimental): Participants will receive one oral dose of psilocybin (capsule), with PAT psychological support and MBCT sessions before, during, and after the psilocybin administration
  Interventions: Combination Product: Psilocybin + MBCT therapy
- Psilocybin with support only (Active Comparator): Participants will receive one oral dose of psilocybin (capsule), with PAT psychological support only sessions before, during, and after the psilocybin administration
  Interventions: Combination Product: Active Comparator: Psilocybin with Support Only

INTERVENTIONS:
Combination Product: Psilocybin + MBCT therapy — The experimental arm has psilocybin with support and MBCT sessions.
  Arms: Psilocybin with support + MBCT
Combination Product: Active Comparator: Psilocybin with Support Only — The active comparator has psilocybin with support only.
  Arms: Psilocybin with support only

SUMMARY:
The goal of this study is to learn how psilocybin delivered with mindfulness-based therapy may help symptoms of posttraumatic stress disorder (PTSD). This is an assessor-blinded, randomized, controlled study in participants with PTSD. The study will investigate the changes in brain activity, connectivity, and microstructural neuroplasticity assessed using EEG/EMG and multimodal MRI measures after administration of one oral dose of psilocybin, accompanied either with standard "psychological support" only; or with standard support plus Mindfulness-based Cognitive Therapy (MBCT).

DETAILED DESCRIPTION:
Many patients with PTSD do not respond or have an incomplete response to treatment with currently available medications that are FDA-approved for PTSD, and/or do not respond to psychotherapies for PTSD. The use of psychedelics (e.g. psilocybin) is being investigated as a new approach to improve symptoms in patients with PTSD and depression, however their mechanism of action is still not well understood. Furthermore, while psychedelics are usually administered in the context of psychological support ("psychedelic assisted therapy", PAT) the kinds of support therapy used and possible interactions with drug with therapy effects is not well understood.

This study will investigate the changes in brain activity, connectivity, and microstructural neuroplasticity, assessed using electroencephalography (EEG) / electromyography (EMG) and functional magnetic resonance imaging (fMRI) /diffusion-weighted magnetic resonance imaging (DWI), after administration of one oral dose of 25 mg synthetic Psilocybin delivered in the context of either non-directive psychological support only (the most common approach for PAT) or in combination with psychological support plus an active form of psychotherapy called Mindfulness-based Cognitive Therapy (MBCT).

Up to 30 participants will be enrolled altogether.

The initial phase of this study will be an open label administration of 25 mg synthetic Psilocybin combined with standard "PAT psychological support" plus MBCT in ten participants with PTSD, to allow us to pilot this new intervention package.

In the next phase of the study, we will randomly assign twenty participants with PTSD into two groups: one group receiving 25 mg of synthetic Psilocybin (open label) combined with standard "PAT support" only, and one group receiving 25 mg of synthetic Psilocybin (open label) combined with standard "support" plus active form MBCT psychotherapy. In both groups, psychological support will be provided before, during and after the administration session. The MBCT group will also receive bi-weekly individual MBCT sessions and will be invited to complete daily homework, as per the MBCT protocol.

Assessments performed at Baseline and on Day 2 and Day 28 after administration will include EEG/EMG, MRI, clinician-administered scales (CAPS-5, MADRS, C-SSRS) and self-report questionnaires to assess PTSD, depression and anxiety symptoms, cognitive testing, self-report questionnaires to evaluate the psychedelic effects of synthetic Psilocybin administration, and blood collection for the Gsα-AC biomarker assay.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is assigned female or male at birth.
2. Participant is aged between 21 to 65 years, inclusive, at Screening.
3. Participant has a BMI of 18 to 35 kg/m2, inclusive, at Screening.
4. Participant is ≥60 kg.
5. Participant has a diagnosis of PTSD (as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-5] established through a clinician interview that includes the Mini-International Neuropsychiatric Interview [MINI]) and CAPS-5.
6. PTSD severity moderate to severe based on CAPS score ≥24.
7. Depression severity moderate to severe based on MADRS score ≥21.

9. Participant has been on a stable dose (no more than 50% change) of antidepressant medication (SSRI) in the last month prior to Screening.

10. Participants capable of producing sperm must use a condom during the trial and for 3 months after their dose of trial medication, if their partner is a person of childbearing potential. In addition, their partner of childbearing potential must use a highly effective method of contraception (i.e., failure rate less than 1% when used consistently and correctly) from dosing until 3 months following dosing.

11. Participants of childbearing potential must agree to use a highly effective method of contraception (i.e., failure rate less than 1% when used consistently and correctly) in combination with use of a condom by a partner who is capable of producing sperm, during the trial and for 3 months after dosing. Such participants must have a negative pregnancy test at Screening and Day 1.

12. Participants of non-childbearing potential who are or were capable of producing eggs (ova) must be postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy or bilateral oophorectomy. Postmenopausal is defined as spontaneous amenorrhea for at least 12 months, and a serum follicle stimulating hormone (FSH) level in the menopausal range, unless the participant is taking hormone replacement therapy or is using hormonal contraception.

13. Provision of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Taking the medications buspirone or venlafaxine in past month
2. Current or previously diagnosed schizophrenia spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, schizotypal disorder, schizophreniform disorder or brief psychotic disorder; current or previous history of bipolar disorder, or current personality disorder (as determined by MINI at Screening).
3. Clinically significant risk of suicidality, as determined through a comprehensive psychiatric interview that incorporates the Columbia Suicide Severity Rating Scale (CSSRS); a score of 4 or higher on the suicidal ideation subscale of C-SSRS (past 6 months) or any suicidal behaviour (lifetime), would be exclusionary.
4. History of substance use disorder within the 12 months, as assessed by a structured clinical interview (Mini International Neuropsychiatric Interview [MINI], Version 7.0.2) or determined by self-report, or intake of >21 units of alcohol weekly, and the inability to refrain from alcohol use from 48 hours before Screening and each scheduled visit until discharge from the study site. One unit is equivalent to a 285 mL glass of full-strength beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.
5. Currently receiving a monoamine oxidase inhibitor, tricyclic antidepressant, other non-SSRI or non-SNRI antidepressants (e.g. bupropion, mirtazapine, etc), an antipsychotic or a mood stabilizer.
6. Exposure to psilocybin, or any other psychedelics, such as ayahuasca, mescaline, LSD or peyote more than 10 times in the last 10 years, or any psychedelic use within 6 months prior to Screening.
7. Use of psychotropic medicine/supplement (or medicine/supplement that would interact with psilocybin) during the 28 days before dosing. Participants may take a stable chronic dose of antidepressant medication(s) and/or sedatives/hypnotics. The Investigator and study team may review medication on a case-by-case basis to determine if its use would compromise participant safety or interfere with study procedures or data interpretation.
8. Family history of schizophrenia or schizoaffective disorder (first degree relatives), or bipolar disorder type 1 (first degree relatives).
9. Clinically relevant history of abnormal physical health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, endocrine, cardiovascular, respiratory, gastrointestinal (including dyspepsia or gastroesophageal reflux disease), hepatic, or renal disorder).
10. Participant has a presence or relevant history of any of the following medical conditions: organic brain disorders (e.g., epilepsy, seizure, intracranial hypertension, intracranial bleed and aneurysmal disease, brain tumor or other medical conditions associated with seizures or convulsions).
11. Diagnosis of hypertension or arrhythmia.
12. Clinically relevant abnormal heart rate (resting supine heart rate >100 bpm) or blood pressure (resting supine systolic blood pressure (SBP) above 140 mmHg or diastolic blood pressure (DBP) above 90 mmHg) at screening. Screening supine SBP, DBP and heart rate for evaluation will be the average of 3 readings obtained after at least 5 minutes rest. Participants with abnormal vital signs which are out of range and deemed clinically significant by the Investigator at Day 1, following triplicate readings.
13. Presence of clinically significant ECG abnormalities at the Screening visit, as defined by medical judgement.
14. QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec at Screening, following triplicate ECG readings.
15. Hypothyroidism and/or current abnormal thyroid function tests. In case of uncertain or questionable screening thyroid function test results, the TSH test may be repeated once during screening. The TSH test must be reviewed to ensure that it is within normal limits before randomizing a participant into the study.
16. Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs, or physical findings at Screening. In case of uncertain or questionable results, tests performed during Screening may be repeated once to confirm eligibility or judged to be clinically irrelevant.
17. Other eligibility considerations (i.e., participant personal circumstances, behavior, and/or any current problem that might interfere with participation or that is incompatible with establishment of rapport or safe exposure to psilocin), as judged by the Investigator.
18. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion (ADME) of the study drug.
19. Any other concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study as outlined in this Protocol, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study.
20. Participant is not fluent in English.
21. Aspartate aminotransferase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT) or total bilirubin levels ≥1.5 x the upper limit of normal (ULN) at Screening. These laboratory evaluations may be repeated once at the discretion of the Investigator. If the repeat test is within the reference range, the participant may be included if the Investigator considers that the previous finding will not introduce additional risk factors.
22. Positive urine test for drugs of abuse or alcohol breath test at Screening or Day 1. A positive test for cannabinoids (e.g., marijuana) at Screening may not exclude a participant if after discussion with and evaluation by the Investigator, the participant agrees not to use any marijuana or other cannabinoid products during the study, and if allowed to participate, the participant must test negative for cannabinoids on Day 1.
23. Participant who consumes excessive amounts of caffeine (e.g., coffee, tea, caffeinated sodas) or (methyl) xanthines (e.g., chocolate) based on the Investigator's determination and discretion.
24. The participant has participated in a clinical study and has received a medication or a new chemical entity within 3 months prior to dosing of current study medication.
25. Known sensitivity to psilocin and/or any excipients present in the formulation. Known fructose malabsorption or intolerance, since the orange drink vehicle for study drug contains fructose.
26. Participant is taking or has taken any drugs known to inhibit monoamine oxidase within 28 days prior to study drug administration.
27. Participant is taking or has taken OTC doses of 5-hydroxytryptophan or St John's Wort within 28 days prior to study drug administration.
28. Strenuous exercise within 48 hours prior to each visit, and while at the study site.
29. Participants capable of producing sperm who will not abstain from sperm donation between first dosing and 3 months after final dosing.
30. Participants of childbearing potential who are pregnant, breastfeeding or planning to conceive.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Changes in parameter estimate of regional brain activity measured by fMRI after one dose of psilocybin in participants with PTSD | Between Baseline and Time point 24 hours and 28 days post-Investigational Product
  Change in Blood oxygenation level dependent (BOLD) fMRI signal after task comparing PAT with MBCT group vs PAT with support only group
Changes in region-to-region connectivity measured by fMRI after PAT with one dose of psilocybin in patients with PTSD | Between Baseline and Time point 24 hours and 28 days post-Investigational Product
  Changes in resting state activity of brain areas comparing PAT with MBCT group vs PAT with support only group
Changes in event related potentials (ERP) after PAT with one dose of psilocybin in participants with PTSD | Between Baseline and Time point 24 hours and 28 days post-Investigational Product.
  Change in ERP as assessed by Electroencephalography (EEG) after task comparing PAT+MBCT group and PAT with support only group
Changes in acoustic startle electromyographic (EMG) response after PAT with one dose of psilocybin in patients with PTSD | Between Baseline and Time point 24 hours and 28 days post-Investigational Product
  Changes in acoustic startle magnitude measured by EMG after task comparing PAT + MBCT group and PAT with support only group

SECONDARY OUTCOMES:
Changes in clinician-assessed PTSD Symptoms after PAT with one dose of psilocybin in patients with PTSD | Baseline to 24 h and 28 days post IP
  Comparison of Clinician Administered PTSD Scale for DSM-5 (CAPS-5 ) score changes from Baseline to 28 days post IP between PAT + MBCT group vs the PAT with support only group. CAPS-5 scores are minimum 0 and maximum 80, higher scores mean a worse outcome
Changes in clinician-assessed Depression Symptoms after PAT with one dose of psilocybin in patients with PTSD | Baseline to 24 hours and 28 days post-Investigational Product (IP)
  Comparison of Montgomery Ashberg Depression Rating Scale (MADRS) score changes from Baseline to 24 hrs and 28 days post IP between PAT + MBCT group vs the PAT with support only group. MADRS scores are minimum 0 and maximum 60, higher scores mean a worse outcome
Changes in Self-report PTSD Symptoms after PAT with one dose of psilocybin in patients with PTSD | Baseline to 24 hrs and 28 days post IP
  Comparison of PTSD Checklist for DSM-5 (PCL-5) score changes from Baseline to 28 days post IP between PAT + MBCT group vs the PAT with support only group. PCL-5 scores are minimum 0 and maximum 80, higher scores mean a worse outcome
Changes in Self-report Depression Symptoms after PAT with one dose of psilocybin in patients with PTSD | Baseline to 24 hrs and 28 days post IP
  Comparison of Beck Depression Inventory - II (BDI-II) score changes from Baseline to 28 days post IP between PAT + MBCT group vs the PAT with support only group. BDI-II scores are minimum 0 and maximum 63, higher scores mean a worse outcome

OTHER OUTCOMES:
Changes in Brain Microstructural Neuroplasticity after PAT with one dose of psilocybin in patients with PTSD | Baseline 24 hours and 28 days post-Investigational Product (IP)
  To assess the role of psychedelic experience on the changes in brain function and/or microstructural neuroplasticity. Correlation between levels of psychedelic experience assessed by self-report questionnaires and the changes in diffusion-weight imagine (DWI) MRI (Neurite Orientation Diffusion and Density)
Proteins and Biomarkers | 24 hours and 28 days post-Investigational Product (IP)
  Correlation between CAPS-5 and MADRS score change and ratio of Gsα, activated to basal adenylyl cyclase (Gsα-AC biomarker score) from Baseline to 24hrs and 21 days post IP between psilocybin with support group vs the psilocybin with active PTSD therapy

IPD SHARING:
Plan to Share IPD: Undecided
We are considering sharing individual participant data sets including all collected IPD, vs all IPD that underlie results in a publication, for the purpose of furthering scientific knowledge